CLINICAL TRIAL: NCT06307522
Title: An Open-Label, Dose-Escalation Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of MRG-001 in Patients With Alcoholic Hepatitis
Brief Title: MRG-001 in Patients With Alcoholic Hepatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedRegen LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MRG24ALC
Record Dates: First submitted 2024-02-26; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Alcoholic Hepatitis; Acute Alcoholic Hepatitis
Keywords: MRG-001; Stem Cells; Immunomodulation; Alcoholic Hepatitis; Hepatitis, Alcoholic; Infection; Liver Diseases, Alcoholic
MeSH Terms: conditions — Hepatitis, Alcoholic; Infections; Liver Diseases, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MRG-001 (0.005 mL/kg) (Experimental): Lowest dose of dose-escalation arm
  Interventions: Drug: MRG-001
- MRG-001 (0.007 mL/kg) (Experimental): Intermediate dose of dose-escalation arm
  Interventions: Drug: MRG-001
- MRG-001 (0.01 mL/kg) (Experimental): High dose of dose-escalation arm
  Interventions: Drug: MRG-001

INTERVENTIONS:
Drug: MRG-001 — Patients will receive subcutaneous administration of MRG-001 at designated visits.

SUMMARY:
The goal of this study is to test MRG-001 (an experimental medication). The purpose of this trial is to assess the dose related safety, Pharmacokinetics, and Pharmacodynamics of MRG-001 in patients with severe alcoholic hepatitis (AH).

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent: Able to provide written informed consent, either personally or through a legally acceptable representative.
2. Male or female patients 21 years of age or older.
3. Onset of jaundice within the prior 8 weeks.
4. Alcohol Consumption: Average daily consumption of more than 40 grams for females or more than 60 grams for males of alcohol for 6 months or longer, with less than 8 weeks of abstinence before the onset of jaundice.
5. Diagnostic Criteria for AH: AH may be diagnosed based on typical serum chemistry or liver biopsy during the current episode of AH, including:

   * Serum bilirubin > 3 mg/dL
   * AST between 50 and 400 IU/L
   * ALT < 400 IU/L
   * AST/ALT ratio > 1.5
6. Maddrey Discriminant Function (MDF): MDF ≥ 32, assuming a control prothrombin time of 12 seconds.
7. Model for End-stage Liver Disease (MELD) Score: MELD score between 21 and 30.
8. Liver Biopsy (Optional): Liver biopsy is not required but may be used to confirm the diagnosis of AH at the Investigator's discretion. If used, the biopsy must have occurred during the current episode.
9. Contraception for Women: Women of childbearing potential must use appropriate birth control throughout the study duration. Contraception for Men: Male patients must agree to use a medically acceptable method of contraception or birth control throughout the study duration.

Exclusion Criteria:

1. Informed Consent: Inability to provide written informed consent, either personally or through a legally acceptable representative.
2. Participation in Other Clinical Trials: Participation in another interventional clinical trial (drug or device) within 30 days of screening and at any time during the study.
3. Concomitant Liver Diseases: Presence of other concomitant causes of liver disease, such as viral hepatitis, autoimmune liver disease, metabolic liver disease, or vascular liver disease.
4. Liver Biopsy Incompatibility: Liver biopsy findings, if conducted, not compatible with alcoholic hepatitis (AH).
5. Absence of Active Infection: No evidence of active infection as determined by the investigator, with specific criteria outlined for diagnosing and treating infections.
6. Uncontrolled Gastrointestinal Bleeding: Presence of uncontrolled gastrointestinal bleeding.
7. History of pre-admission refractory ascites, as defined by the frequency of paracenteses despite diuretic therapy.
8. Significant pre-existing organ dysfunction in various systems, including lung, heart, kidney, hematologic, neurological, and spleen-related conditions.

   1. Lung: Receiving supplemental home oxygen therapy at baseline for pre-existing medical condition (other than COVID-19), as documented in medical record.
   2. Heart: Pre-existing congestive heart failure defined as an ejection fraction <20% as documented in the medical record. Clinically significant ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation), unstable angina, myocardial infarction (past 3 months), heart and coronary vessel surgery (past 3 months), significant valvular heart disease, uncontrolled arterial hypertension with systolic blood pressure >180 mm Hg and diastolic blood pressure >110 mm Hg.
   3. Renal: End-stage renal disease requiring renal replacement therapy or creatintine clearance <30 mL/min.
   4. Hematologic: Baseline platelet count <30,000/mm3 or hemoglobin levels <6.0 g/dL.
   5. Neurological: Stage ≥3 hepatic encephalopathy by West Haven criteria.
   6. History of splenectomy or splenomegaly (spleen weighing > 750 g).
9. Presence of any active malignancy or malignancy diagnosed within the last five years, excluding curable skin cancer.
10. Patients requiring the use of vasopressors or inotropic support, excluding stabilized conditions within the first 7 days of hospital admission.
11. Presence of co-infection with human immunodeficiency virus (HIV) or active tuberculosis on chest X-ray at study entry.
12. History of organ or bone marrow transplantation, excluding corneal transplant, or recent chronic use of immunosuppressive drugs.
13. Positive urine drug screen for specific substances, excluding THC and prescription medications.
14. Hypersensitivity to either of the components of MRG-001.
15. If female, known pregnancy, positive serum pregnancy test, or lactating/breastfeeding.
16. Underlying diseases that might be complicated or exacerbated by proposed treatments or confound assessment of study drug, as determined by the site investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Treatment-Emergent Adverse Events | 28 Days
  Assess the safety and tolerability of MRG-001 in patients with alcoholic hepatitis (AH) as determined by the absence of suspected unexpected serious adverse reaction (SUSAR).

SECONDARY OUTCOMES:
Pharmacokinetic Response | 28 Days
  Determine the pharmacokinetics (PK) of MRG-001 in patients with AH. Trough levels (Ctrough) of plerixafor and tacrolimus will be measured throughout the study.
Pharmacodynamic Response | 28 Days
  The PD response will be measured by flow cytometry. The absolute number of CD34+ hematopoietic stem cells in the peripheral circulation will be assessed and compared to baseline levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ali R Ahmadi, MD PhD, Study Director — MedRegen LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahmadi AR, Atiee G, Chapman B, Reynolds L, Sun J, Cameron AM, Wesson RN, Burdick JF, Sun Z. A phase I, first-in-human study to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of MRG-001 in healthy subjects. Cell Rep Med. 2023 Sep 19;4(9):101169. doi: 10.1016/j.xcrm.2023.101169. Epub 2023 Aug 25. PMID 37633275
- See also: Company Profile — http://medregenco.com